CLINICAL TRIAL: NCT07181525
Title: Construction and Validation of a Predictive Model for the Efficacy of Different Biologics in Inflammatory Bowel Disease
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dai Yun, Professor, Peking University First Hospital
Other Study IDs: 2025R0267-0001
Record Dates: First submitted 2025-08-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Inflamatory Bowel Disease
Keywords: inflammatory bowel disease; machine learning; biologics
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAT group: IBD patients treated with cytokine antagonists
  Interventions: Drug: anti-cytokine antibodies
- IAT group: IBD patients treated with integrin antagonists
  Interventions: Drug: anti-integrin antibodies

INTERVENTIONS:
Drug: anti-cytokine antibodies — Different kinds of biologics used to treat inflammatory bowel disease (including anti-cytokine antibodies)
  Groups: CAT group
Drug: anti-integrin antibodies — Different kinds of biologics used to treat inflammatory bowel disease (including anti-integrin antibodies)
  Groups: IAT group

SUMMARY:
Inflammatory bowel disease (IBD) is a group of chronic progressive gastrointestinal diseases that can recur throughout life and for which there is no cure. Biologics, the first line of treatment, are not only expensive, but also 30-50% of patients lack response to this type of drug therapy. However, there is a lack of reliable methods to predict the clinical efficacy of biologics. The aim of this study is to construct a reliable model to predict patients' response to biologics therapy by comprehensively analysing patients' clinical characteristics, biomarkers and other information to guide individualized therapy. In this study, we will collect clinical data from IBD patients at Peking University First Hospital, including but not limited to patients' baseline characteristics, biomarker levels, and efficacy responses, etc. We will establish a complete patient dataset using a cohort study, train and test the dataset by applying correlation analysis, multiple regression analysis, and machine learning algorithms (e.g. neural networks etc), establish and compare the prediction effects of different models The optimal model is selected for encapsulation and developed into a user-friendly clinical prediction tool. This study will contribute to clinical decision making for IBD patients, improve treatment outcomes, and reduce unnecessary healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically diagnosed with IBD in our hospital
* Disease activity is in the active stage
* Receiving biologics after diagnosis
* Have relevant data on clinical evaluation results after receiving biologics treatment

Exclusion Criteria:

* IBD patients who have not been treated with biologics after diagnosis
* Patients diagnosed with IBD but also with other autoimmune diseases that require biologics to be treated
* Patients with hematological diseases and other systemic chronic inflammatory diseases involving the intestine Patients with serious complications including malignant tumors and gastrointestinal perforation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult inflammatory bowel disease patients in our hospital have no specific selection such as race, gender, or age.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
disease activity | up to 8 weeks
  For UC patients, the modified Mayo scoring system was used to evaluate the disease activity of UC patients, and the items involved in the score included the number of bowel movements, blood in the stool, endoscopic performance and physician's overall evaluation, and the sum of the scores was <2 points without a single sub->1 is considered to be in remission, ≥ 3 points or a single sub-item> 2 points are considered active period; For CD patients, the severity of disease activity is assessed using Best's Crohn's disease activity index (CDAI), including the number of loose stools, abdominal pain, general conditions, extraintestinal manifestations and complications, opioid antidiarrheal use, abdominal masses, decreased hematocrit, and weight loss≥<.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided